CLINICAL TRIAL: NCT06113705
Title: Imaging and Biological Markers for Prediction and Identification of Glioblastoma Pseudoprogression: a Prospective Study.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Mediolanum Cardio Research (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Research Administrator Manager, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NEURAD-2022-001
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Multidisciplinary and innovative approach based on plasma markers of inflammation (cytokines, circulating RNA, and extracellular microvesicles), and multimodal imaging using 18F-GE-180 positron emission tomography (PET) and advanced MRI techniques,
  Interventions: Diagnostic Test: 18F-GE-180 PET; Diagnostic Test: Advanced MRI; Other: Collection of hematopoietic stem cells; Other: Blood withdrawal; Other: Collection of Cancer Stem Cells

INTERVENTIONS:
Diagnostic Test: 18F-GE-180 PET — PET examination of glioblastoma using 18F-GE-180 PET radio-metabolic marker
Diagnostic Test: Advanced MRI — MRI examination using advanced sequences to characterize tumor microstructure and function
Other: Collection of hematopoietic stem cells — Hematopoietic stem cells will be collected by the aspiration of bone marrow during the surgical intervention for tumor resection
Other: Blood withdrawal — blood withdrawal for evaluation of plasma biomarkers of inflammation, circulating microvesicles, and RNA
Other: Collection of Cancer Stem Cells — Glioblastoma stem cells (GSCs) will be isolated from the tumor

SUMMARY:
The goal of this interventional study is the development and validation of imaging markers, MRI and PET, plasma biomarkers, and/or cell markers that could support clinicians and researchers in differentiating pseudoprogression from true tumor progression in routine clinical activities and clinical trials in patients affected by glioblastoma.

The endpoints of the study are:

* the elaboration of predictive models using imaging advanced biomarkers, PET and MRI, biological serum markers, and cancer cell derived makers to differentiate tumor pseudoprogression or real progression in patients affected by glioblastoma who underwent therapeutical protocol as per treating physicians' indications (Stupp or hypofractionated RT)
* to establish an in vivo murine model of pseudoprogression by orthotopic transplantation of glioblastoma stem cells derived from thirty-five patient subjected to subsequent treatment with irradiation and temozolomide administration.

Participants will undergo:

* baseline MRI and 18F-GE-180 PET imaging, and blood withdrawal
* surgery
* collection of glioblastoma stem cells (and hematopoietic stem cells from a sub-group of subjects)
* standard treatment with radiotherapy and chemotherapy
* MRI every 3 months
* PET and blood withdrawal in case of MRI evidence of either suspected tumor progression or pseudoprogression
* second surgery OR stereotactic biopsy OR clinico-radiological follow-up as for standard of care according to the Institutional Multidisciplinary Brain Tumor Board

DETAILED DESCRIPTION:
Rationale

Glioblastoma (GBM) is the most common malignant primary tumor of the central nervous system characterized by an extremely severe prognosis with a median survival of 14-16 months from diagnosis. Patients affected by high-grade gliomas are treated with a combination of radiotherapy and temozolomide chemotherapy. To date, the efficacy of the treatment is assessed through MRI which shows evidence of early radiological progression in up to 50% of all patients. Importantly, signs of tumor progression on MRI images may actually represent pseudoprogression in up to 64% of cases meaning that within 6 months from the end of the radiation treatment 20-30% of patients show increased contrast enhancement that resolves on subsequent MRI scans without changes in the treatment. Pseudoprogression is a phenomenon likely related to inflammation and disruption of the blood-brain barrier (BBB) caused by radiation and by the concurrent temozolomide treatment. Being a self-resolving consequence of the therapy rather than a sign of tumor growth, mistaking pseudoprogression for real progression leads to premature discontinuation of therapy and inappropriate evaluation of progression free survival and response rate in clinical trials impairing clinical practice.

Therefore, the differentiation of pseudoprogression from true progression is both a challenge in everyday clinical activity and a relevant problem in clinical trials and research.

A major limitation to the development and assessment of efficacy of current and new therapies in the setting of brain tumors, both at preclinical and clinical levels, however, is the lack of reliable trial endpoints.

A combination of advanced imaging methods, MRI and PET, with innovative techniques investigating cancer-specific biology will allow a holistic characterization of the tumor from multiple aspects crucial to enable a personalized diagnostic and therapeutical approach.

Objective

The main goal of the project is the development and validation of imaging markers, MRI and PET, plasma biomarkers, and/or cell markers that could support clinicians and researchers in differentiating pseudoprogression from true tumor progression in routine clinical activities and clinical trials in patients affected by GBM.

Main trial endpoints

The primary endpoint of the study is the elaboration of predictive models (evaluation of specificity and sensitivity) using imaging advanced biomarkers, PET and MRI, biological serum markers, and cancer cell derived makers to differentiate tumor pseudoprogression or real progression in patients affected by GBM who underwent therapeutical protocol as per treating physicians' indications (Stupp or hypofractionated RT).

Secondary trial endpoints

We aim to establish an in vivo murine model of pseudoprogression by orthotopic transplantation of GSCs derived from thirty-five patient subjected to subsequent treatment with irradiation and temozolomide administration.

Trial design

This is a pilot prospective interventional clinical trial using a novel 18F-GE-180 PET radio-metabolic marker (AxMP) and MRI with advanced sequences with no modification of standard of care treatment and additional diagnostic procedures that do not pose more than minimal additional risk or burden to the subjects compared to normal clinical practice. The trial will enroll 75 patients in 42 months and will be concluded in 60 months.

Trial population

The trial will prospectively enroll 75 patients affected by isocitrate dehydrogenase gene (IDH)-wild type Glioblastoma, with an age above 18 years old , who will undergo standard of care treatment.

Interventions

Before surgery and starting the standard treatment with RT and chemotherapy, all subjects will undergo baseline MRI and 18F-GE-180 PET imaging, and blood withdrawal for evaluation of plasma biomarkers of inflammation, circulating microvesicles, and RNA. MRI exams will then be performed as per standard practice of care every 3 months and in case of clinical deterioration suggesting possible disease recurrence/progression. A second PET-scan along with plasma sample collection will be performed only in case of MRI evidence of either suspected tumor progression or pseudoprogression. In case of MRI evidence of an increase in tumor size (either suspected true tumor progression or pseudoprogression), as for standard of care, the Institutional Multidisciplinary Brain Tumor Board (composed of neurosurgeons, neuro-oncologists, neuroradiologists, radiotherapists) will discuss each patient for determining clinical indication and feasibility of second surgery. In those patients in whom second surgery is not indicated, a stereotactic biopsy will be considered if feasible, safe, and clinically useful. If a stereotactic biopsy is not feasible and safe, a 3-month follow-up will be planned before a change in treatment. When available, pathology will be considered as the gold standard for differentiation pseudoprogression from true tumor progression. In all other subjects, follow-up and overall survival data will be evaluated for this differentiation. In all the subjects, overall survival data will be also recorded for statistical analyses.

Cancer Stem Cells /CSC) will be collected form 35 patients and Hematopoietic Stem Cells (HSC) from 10 patients for the creation of a vitro and in vivo murine model.

Ethical considerations relating to the clinical trial including the expected benefit to the individual subject or group of patients represented by the trial subjects as well as the nature and extent of burden and risks This trial will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki and International Conference on Harmonization Good Clinical Practice guideline as well as international and national legal and regulatory requirements.

All study participants will receive the standards of care for GBM. The additional diagnostic procedures (PET scan with a novel tracer and high resolution 3 Tesla scanner MRI) do not entail specific risks for the patient. At every time point (at least before surgery, before RT and in case of pseudoprogression) additional blood samples for the determinations of markers of inflammation and the isolation of circulating microvesicles and RNA will be collected from the patients. Glioblastoma stem cells will be isolated from the tumoral mass excised during glioblastoma surgery in 35 patients; hematopoietic stem cells will be obtained from 10 consenting patients at the time of surgery by aspiration of 30-40ml of bone marrow from the iliac crests, as per standard clinical practice. Since the biopsy will be performed under general anesthesia, the patient should not experience discomfort.

There are no expected benefits for the individual patient, but the study results might provide important advances for the treatment of future patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sex and any race age >= 18.
2. Histologically proven glioblastoma multiforme wild type for IDH1-2 mutation with MGMT promoter methylated or unmethylated OR subjects with medical history, clinical sign and symptoms and MRI findings highly consistent with the diagnosis of IDH wild type glioblastoma.
3. Patient eligible to undergo treatment with TMZ and RT (Stupp protocol or hypofractionated protocol as per Institutional Multidisciplinary Brain Tumor Board's decision)
4. Willingness and ability to sign the informed consent and participate to the trial.

Exclusion Criteria:

1. Patient age <18.
2. Patient not eligible to undergo treatment with TMZ and RT (Stupp protocol or hypofractionated protocol as per Institutional Multidisciplinary Brain Tumor Board's decision).
3. Patient presenting contraindication to undergo contrast-enhanced MRI (pacemaker or allergy to gadolinium).
4. Patient HIV1-2 positive.
5. Patient affected by other systemic infective or inflammatory diseases or involving the central nervous system (multiple sclerosis, lupus, Chron, rheumatoid arthritis).
6. Patients that are pregnant or breast-feeding. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive models of pseudoprogression | From baseline assessment to the last visit of the patient as per protocol
  predictive models (evaluation of specificity and sensitivity) using imaging advanced biomarkers, PET and MRI, biological serum markers, and cancer cell derived makers to differentiate tumor pseudoprogression or real progression in patients affected by GBM who underwent therapeutical protocol as per treating physicians' indications (Stupp or hypofractionated RT)

SECONDARY OUTCOMES:
Glioblastoma Stem Cells (GSCs) isolation and in vitro model | starting from the day of the first surgery
  Glioblastoma stem cells (GSCs) will be isolated from the tumors of the patients enrolled, characterized at the molecular and functional level before and after in vitro treatment with radiations and TMZ, to identify candidate cellular phenotypes and molecular pathways possibly associated with pseudoprogression

OTHER OUTCOMES:
Glioblastoma and Hematopoietic Stem Cells isolation and in vivo model | Starting from the day of the first surgery
  To establish and characterize in vivo murine models of pseudoprogression by orthotopic transplantation of patient-derived GSCs in nonobese diabetic scid gamma (NSG) mice previously repopulated with individual patients' hematopoietic stem and progenitor cells to reproduce a humanized environment and to correlate in vivo imaging findings and plasma markers with pathology

CONTACTS AND LOCATIONS:
Overall Officials: Letterio S Politi, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- IRCCS Istituto Clinico Humanitas, Rozzano, Italy